CLINICAL TRIAL: NCT03928769
Title: Role of Telomere Length in Arterial Smooth Muscle Cells and Circulating/Tissue Endothelial Progenitors in the Development of Atherosclerotic Lesions: Set up of the Experimental Model
Brief Title: PROGENitors, TELomeres and ARTerial Aging
Acronym: PROGENTELART
Status: Suspended | Type: Observational
Why Stopped: Covid-19 Pandemics
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A00143-54
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-01

CONDITIONS: Atherosclerosis of Artery
Keywords: Telomere length; Endothelial progenitor cell; Smooth muscle cell; Senescence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Patients with traumatic vascular injury, ultimately corresponding to control patients
- Atheroma Group: Patients will be included either in the atheromatous group (patients with atheromatous pathology) or in the control group (patients without atheromatous pathology), according to the clinical evaluation.
  In the atheromatous group, subjects must have a clinically significant atheromatous pathology.
  The investigator must specify the site (s) affected by the atheroma: carotid artery, coronary artery, aorta, renal artery, mesenteric artery or lower limb artery.

SUMMARY:
The prevailing view in telomere epidemiology is that leukocyte telomere length (LTL) is associated with atherosclerotic cardiovascular disease (ACVD) since it serves as a biomarker of the cumulative burden of inflammation and oxidative stress during adult life. However, our recent results indicate that telomere length (TL) is mainly determined before adulthood, by TL at birth and TL attrition during growth. They also demonstrate that short telomeres precede the clinical manifestation of atherosclerosis. The investigators therefore hypothesize that LT is not a simple marker, but a major determinant of arterial aging.

Two mechanistic hypotheses may explain an active role of short telomeres in accelerated arterial aging and development of ACVD.

The first is that a short TL at the leukocyte level reflects a short TL in endothelial progenitor cells (EPC). Cell replicative capacity being TL-dependent, short telomeres in the EPC would therefore be responsible for diminished replication capacity and vascular repair potential, thereby increasing the vulnerability for developing age-related arterial diseases.

The second hypothesis is that a short LTL reflects short TL in arterial wall cells, leading to an increase in the number of senescent vascular cells. Senescent cells are known to alter their secretion pattern, a phenomenon called senescence-associated secretory phenotype (SASP), and thus contribute to tissue injury by promoting inflammation and tissue remodeling leading to lesion progression.

These assumptions cannot be tested by LTL measurements alone. The investigators propose, therefore, a model that makes it possible to examine different elements of TL dynamics in different tissues and cell types: leukocytes, circulating EPCs, in situ EPCs and arterial resident cells (mainly smooth muscle cells) in patients with or without atherosclerosis.

Our model is based on the following observations:

* TL is synchronized (equivalent) across somatic tissues/cells of the newborn: an individual with short telomeres (relative to his pairs) in one tissue should also have short telomeres (relative to his pairs) in other tissues.
* TL in EPCs (both circulating and in situ) determines the cell proliferative ability and therefore capacity for vessels repair during aging.
* TL in the cells of the arterial wall determines the number of senescent cells that therefore contribute to tissue injury through their change of phenotype.

The general aim of the present project is to examine the mechanistic links between arterial aging and TL in these different cell types.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* Patient for whom a vascular surgery is programmed, and whose nature allows obtaining of arterial segment without any harm for the health of the patient
* Patient for whom a blood sample is planned on the day of the procedure
* Person who has received complete information on the organization of the research and who has not objected to his participation and the exploitation of his data
* Compulsory affiliation to social security

Exclusion Criteria:

* Patient who has previously undergone radiotherapy at the sampling site
* Patient with cancer at the sampling site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment is expected in patients undergoing surgery giving access to arterial surgical residues.
  Recruiter Service: Vascular Surgery at Nancy-Brabois University Hospital (Prof. Serguei Malikov)
  As part of the clinical care, the samples available according to the groups are as follows:
  * for the group suffering from atheromatous pathology: lesion (pathological zone) and lesion border (healthy zone)
  * for the group with traumatic vascular injury: lesion (but non-atheromatous lesion, therefore considered as control) and lesion border.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-04-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Circulating EPC levels | Inclusion visit
  Circulating EPC levels measured from whole blood specimens after primary culture of peripheral blood mononuclear cells (PBMC) on fibronectin (in cells per million of PBMCs)
Tissue EPC levels | Inclusion visit
  Tissue EPC levels measured from arterial wall cells in healthy and pathological zones obtained after enzymatic digestion, cell sorting and primary culture.

SECONDARY OUTCOMES:
TL in EPC | Inclusion visit
  Description and comparison of telomere lengths in circulating and tissue endothelial progenitors in patients with atheromatous pathology and those with traumatic vascular disease.
  The telomere length in the different cell types (expressed in kb) will be measured by Southern blot after DNA extraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided